CLINICAL TRIAL: NCT05209802
Title: High-intensity Aquatic Exercise for Adults with Rheumatic Diseases (AquaHigh)
Brief Title: High-intensity Aquatic Exercise for Adults with Rheumatic Diseases
Acronym: AquaHigh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: The Dam Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 272749
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-07

CONDITIONS: Rheumatic Diseases
Keywords: Rheumatic Diseases; Aquatic exercise; High-intensity
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Exercise (Experimental): High intensity interval exercise training (4 x 4 minutes of intensity above 17 on the Borg Rating of Perceived Exertion)
  Interventions: Other: Group A: High intensity exercise training
- B: Exercise (Active Comparator): Moderate intensity exercise training
  Interventions: Other: Group B: moderate intensity exercise training

INTERVENTIONS:
Other: Group A: High intensity exercise training — Both group will receive aquatic exercise training twice a week for 12 weeks at different intensities
  Arms: A: Exercise
Other: Group B: moderate intensity exercise training — Both group will receive aquatic exercise training twice a week for 12 weeks at different intensities
  Arms: B: Exercise

SUMMARY:
The purpose of this study is to compare aquatic high intensity interval training with moderate intensity exercise training on exercise capacity in a population with rheumatic diseases.

DETAILED DESCRIPTION:
Exercise is important to manage rheumatic diseases (RDs). In 2007, the American College of Sports Medicine (ACSM) launched a global initiative to advocate the use of exercise not only to prevent illness but to serve as a key element in the management and treatment of multiple chronic diseases. Their "Exercise is Medicine" initiative promotes exercise as a highly potent free medicine with few side effects. Despite catchphrases such as "best drug ever," few adhere to the global recommendations for weekly physical activities. Exercise is one of the therapeutic strategies that helps minimise deleterious effects on the musculoskeletal system generated by aging while preserving independence, promoting weight control, and maintaining or improving quality of life, functional capacity, and emotional well-being. However, exercises performed on the ground can aggravate joint pain and increase the risk of falls among those with RDs. Aquatic exercises are a popular adjunct treatment modality for patients with inflammatory RDs. Aquatic exercises are highly preferred by people with RDs, who are more likely to report feeling better than those treated with similar exercises on land. A preference for a water-based rehabilitation or environment may enable greater exercise compliance.

A systematic review and meta-analysis from 2011 concluded that the effects of aquatic exercise for adults with arthritis appears comparable to land-based exercise. When people are unable to exercise on land or find it difficult, aquatic programs provide an enabling alternative strategy.

Aquatic exercise programmes have been criticised for being non-progressive or low-intensive. One possible advantage of the aquatic environment is that the people with chronic diseases may be able to train at higher intensities than on land.

The effectiveness of aquatic exercise needs further comprehensive investigation, particularly related to the link between load, types of exercise, and degree of changes in physical functioning and physical fitness.

Method:

* Design: The study will be a randomized clinical trial. Patients will be recruited from different municipalities in Norway with possibilities of pool training in temperate water (between 30-34°C to be optimal).
* Intervention group: The intervention group will receive aquatic high intensity interval exercise training twice a week for 12 weeks.
* Control group: The control group will receive aquatic moderate intensity exercise training twice a week for 12 weeks.
* Sample Size Estimation: Sample size is calculated on the basis of the primary outcome variable, where a between-group difference in VO2peak of 15% or 3.5 mL∙kg-1∙min-1 is considered to be of clinical relevance. Both groups are receiving an exercise intervention, therefore we estimate a smaller between group difference to be 2.0 mL∙kg-1∙min-1. Using a reported standard deviation of change in VO2peak of 3 and 80% power to detect this difference, approximately 35 participants are required in each group. To allow for a possible 20% drop-out rate, we plan to randomise 84 patients in total (i.e. 42 per group).
* Statistical analyzes: Descriptive data are reported for variables of interest and will be analysed following the intention-to-treat principle. Prospective differences in primary and secondary outcomes and baseline characteristics between the intervention group and the control group will be assessed by t-tests for continuous and normal distributed variables and non-parametric tests for categorical variables. Multiple linear regression modelling is used to control for confounding differences between study groups.

The study will provide evidence-based knowledge for performing high-Intensity water workout in municipalities and investigates the factors that determine successful effects on physical fitness, disease activity and pain and tests the programme's utility for municipal health care services.

ELIGIBILITY:
Inclusion Criteria:

Individuals who

* are 18 years or older,
* have a diagnosis of any kind of RDs,
* can walk with or without a walking aid and
* understand Norwegian.

Exclusion Criteria:

* medical contraindications to high intensity exercise,
* life expectancy below 1 year and
* currently participating or have participated in aquatic high intensity exercise programs or trials during the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption | Change from baseline at 3 and 6 months
  Physical capacity will be assessed with a maximal walking treadmill test for estimation of peak oxygen consumption. A modified Balke protocol on a treadmill will be used.

SECONDARY OUTCOMES:
Change in 30 STS | Change from baseline at 3 and 6 months
  The 30 sec sit-to-stand test (30STS) will be used is a measure of lower extremity strength
Change in Patients Global Assessment score | Change from baseline at 3 and 6 months
  Change in Patients Global Assessment score (PGA) is a self-reported measure in which the patient's overall disease activity is measured. The phrasing of PGA is not standardized, but the PGA of the American College of Rheumatology (ACR) and EULAR is based on the question "In all the ways in which your RDs affect you, how would you rate the way you felt over the past week?" PGA is reported on a 100-mm Visual Analogue Scale (VAS). Higher scores represent a high level of disease activity. PGA is reliable for the assessment of both joint and skin disease and a PGA score < 20 is defined as low disease activity.
Change in the 8-item Patient-Reported Outcomes Measurement Information System (PROMIS) physical function form (PF-8a). | Change from baseline at 3 and 6 months
  The 8-item Patient-Reported Outcomes Measurement Information System, (PROMIS) physical function form (PF-8a) is a brief patient-reported measure of physical function, Scale 5 (best) to 1 (worst)
Change in Quality of Life | Change from baseline at 3 and 6 months
  Euro Quality of life questionnaire (EQ5D-5L), Scale 1 (best) to 5 (worst) and Scale 0 (worst) to 100 (best)
Change in patients' level of physical activity | Change from baseline at 3 and 6 months
  The University of California, Los Angeles (UCLA) Activity Scale measures the patients' level of physical activity on a 10-point scale based on 10 descriptive activity levels ranging from wholly inactive and dependent to regular participation in impact sports. Scale 1 (worst) to 10 (best)
Change in reported pain | Change from baseline at 3 and 6 months
  The Numeric Rating Scale (NRS) for pain will be measured at rest and in activity on a 0-10 NRS. The patients mark a number from 0 (no pain) to 10 (worst pain)
Change in fatigue | Change from baseline at 3 and 6 months
  The Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF-MDQ) score assesses NRS for fatigue severity, effect, and coping during the past 7 days. All three dimensions are rated from 0-10, and the total score is obtained by dividing the sum of individual scores by 3
Demographic variables | Baseline and change from baseline to 3 and 6 months for age, smoking, medications
  We will record the following variables: age, living alone (yes/no), BMI, educational level, smoking (yes/no), medications, taking analgesics (yes/no), and comorbidities.
Training diary | From baseline to 3 months. From 3 to 6 months is optional
  Exercise frequency Participants are asked to record group-based exercise sessions and other individual exercise sessions in a training diary.
  Exercise intensity Participants are asked to record group-based exercise sessions in a training diary. Exercise intensity is recorded by use of a Borg RPE scale.
  Session deviation Participants are asked to record group-based exercise session in a training diary. Participants are asked to recording both early session terminations and absences from scheduled training sessions.
  Exercise-related adverse events Participants are asked to record group-based exercise session in a training diary. Participants are asked to record exercise-related adverse events.
Self-reported physical activity (HUNT) | From baseline to 3 months and 6 months
  Average frequency (never/<1 per week/1 per week/2-3 per week/almost every day), intensity (easy without losing my breath or breaking into a sweat/so hard that I lose my breath and break into a sweat/I push myself to near-exhaustion) and duration (less than 15 minutes/15-29 minutes/30 minutes to 1 hour/more than 1 hour) of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Bunæs-Næss, MSc, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metroplitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bunaes-Naess H, Nilsson BB, Kvael LAH, Heywood SE, Gerritsen RB, Heiberg KE. Effects of aquatic high-intensity interval training on patient-reported outcome measures and quality-adjusted life-years in adults with rheumatic and musculoskeletal diseases: a secondary analysis of the AquaHigh randomised controlled trial. BMJ Open. 2025 Nov 13;15(11):e102841. doi: 10.1136/bmjopen-2025-102841. PMID 41238358
- [Derived] Bunaes-Naess H, Heywood SE, Kvael LAH, Heiberg KE, Nilsson BB. Effects of aquatic high-intensity interval training on aerobic capacity in adults with rheumatic and musculoskeletal diseases: the AquaHigh randomised controlled trial. BMJ Open. 2025 Mar 24;15(3):e090612. doi: 10.1136/bmjopen-2024-090612. PMID 40132852